CLINICAL TRIAL: NCT06996730
Title: A Double-Blind, Placebo-Controlled, Double-Dummy Study of Donanemab and RG6289 in PSEN1 E280A Mutation Carriers, and in Non-Randomized, Placebo-Treated Non-Carriers From the Same Kindred, to Evaluate the Efficacy and Safety of Donanemab, RG6289, or the Combination of Donanemab and RG6289, in the Treatment of Autosomal-Dominant Alzheimer's Disease
Brief Title: A Study of Donanemab, RG6289, or the Combination of Donanemab and RG6289 in Presenilin 1 (PSEN1) E280A Mutation Carriers for the Treatment of Autosomal-Dominant Alzheimer's Disease
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Banner Health (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Universidad de Antioquia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: API-2; 1R01AG086363-01 (NIH)
Record Dates: First submitted 2025-04-29; First posted 2025-05-30 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Autosomal Dominant Alzheimers Disease; Early Onset Alzheimer Disease; Alzheimers Disease
Keywords: Dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — donanemab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Part 1: Donanemab (Experimental): Donanemab will be administered per the schedule specified in the treatment arm for all PSEN1 E280A Carriers
  Interventions: Drug: Donanemab
- Part 1: Donanemab placebo (Placebo Comparator): Donanemab placebo will be administered per the schedule specified in the treatment arm for all PSEN1 E280A Non-Carriers
  Interventions: Drug: Donanemab placebo
- Part 2: Donanemab + RG6289 placebo (Experimental): Donanemab plus RG6289 placebo will be administered per the schedule specified in the treatment arm for all PSEN1 E280A Carriers
  Interventions: Drug: Donanemab; Drug: RG6289 placebo
- Part 2: RG6289 + Donanemab placebo (Experimental): RG6289 plus donanemab placebo will be administered per the schedule specified in the treatment arm for all PSEN1 E280A Carriers
  Interventions: Drug: RG6289; Drug: Donanemab placebo
- Part 2: RG6289 plus donanemab (Experimental): RG6289 plus donanemab will be administered per the schedule specified in the treatment arm for all PSEN1 E280A Carriers
  Interventions: Drug: Donanemab; Drug: RG6289
- Part 2: RG6289 placebo plus donanemab placebo (Placebo Comparator): RG6289 placebo plus donanemab placebo will be administered per the schedule specified in the treatment arm for all assigned PSEN1 E280A Carriers and all PSEN1 E280A Non-Carriers
  Interventions: Drug: Donanemab placebo; Drug: RG6289 placebo

INTERVENTIONS:
Drug: Donanemab — IV Infusion
  Arms: Part 1: Donanemab; Part 2: Donanemab + RG6289 placebo; Part 2: RG6289 plus donanemab
Drug: RG6289 — Oral tablet
  Arms: Part 2: RG6289 + Donanemab placebo; Part 2: RG6289 plus donanemab
Drug: Donanemab placebo — IV placebo
  Arms: Part 1: Donanemab placebo; Part 2: RG6289 + Donanemab placebo; Part 2: RG6289 placebo plus donanemab placebo
Drug: RG6289 placebo — Oral tablet placebo
  Arms: Part 2: Donanemab + RG6289 placebo; Part 2: RG6289 placebo plus donanemab placebo

SUMMARY:
The study will be conducted in 2 blinded parts (Part 1 and Part 2). In Part 1, study participants who are mutation carriers will receive active donanemab and non-mutation carriers will receive placebo-donanemab for up to 18 months (76 weeks), with a minimum treatment period of 9 months. Amyloid PET scans will be conducted at screening, 9, and 18 months in Part 1. Participants who are at or below 11 CL at screening or reach complete amyloid plaque clearance as measured by florbetapir F18 PET (defined as ≤11 CL) at 9 months will initiate Part 2. Participants who are ≤11 CL at screening may delay their entry into Part 2 for up to 6 months at the discretion of the Investigator. All remaining participants will start Part 2 after completing 18 months (76 weeks) in Part 1 independent of amyloid results. Non-carriers will receive placebo in both Parts 1 and 2.

In Part 2, study participants who are mutation carriers will be randomized 1:1:1:1 in a full factorial design to receive either RG6289 + placebo-donanemab (RG6289 alone group), donanemab + placebo-RG6289 (donanemab alone group), the combination of RG6289 and donanemab (combination group), or placebo-RG6289 and placebo-donanemab (placebo group). All non-carriers will be assigned to the placebo group. CDR-GS at the end of Part 1 and the amyloid level using the last completed amyloid PET scan in Part 1 will be used for stratification. All study participants will participate in a double-dummy design for the duration of Part 2 receiving both an intravenous (IV) infusion at the required interval for the donanemab or matching placebo as well as a daily oral treatment of RG6289 or matching placebo.

An exploratory outcome of Part 1 is a comparison of the amyloid clearance between this ADAD cohort and historical controls using propensity score matching. The primary outcome in Part 2 is change from the start of Part 2 through the end of Part 2 in brain amyloid load in PSEN1 E280A mutation carriers as measured by amyloid PET imaging. Other endpoints will include fluid and imaging biomarkers and measures of cognition and functioning. The maximum study duration for any individual participant will be 3 years, not including the screening or follow-up periods

ELIGIBILITY:
Inclusion Criteria:

* Membership in PSEN1 E280A mutation carrier kindred.
* Agrees to conditions of, and is willing to undergo, genetic testing (e.g., APOE, PSEN1 E280A, and other genetic testing allowed by local regulatory requirements).
* Males and females aged 25-65 inclusive.
* Must meet one of the following criteria:

  a. Determined to be cognitively normal as defined by an MMSE of ≥24 for participants with less than 9 years of education or MMSE of ≥26 for participants with 9 or more years of education. b. Or determined to have MCI with amnestic presentation as defined by:

  1. Cognitive concern in the judgment of the Investigator, based in part on the: i. CERAD Word List: Recall <3 for participants with less than 9 years of education. ii. CERAD Word List: Recall <5 for participants with 9 or more years of education. iii. Preservation of independence in functional activities in the judgment of the Investigator. c. Or determined to have mild AD dementia as defined by:
  1. Meets the 2011 National Institute on Aging and the Alzheimer's Association (NIA-AA) criteria for probable AD, and
  2. Has a CDR-GS of 0.5 or 1, with the memory box score ≥0.5.

     Exclusion Criteria:
* Significant medical, psychiatric, or other neurological condition or disorder documented by history, physical, neurological, laboratory examinations that would place the participant at undue risk in the Investigator's judgment or impact the interpretation of efficacy.
* History of stroke.
* History of severe, clinically significant (persistent neurological deficit or structural brain damage) CNS trauma (e.g., cerebral contusion).
* Current presence of bipolar disorder or other clinically significant major psychiatric disorder according to Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, Text Revision (DSM-5-TR) or symptom (e.g., hallucinations, agitation, paranoia) that could affect the participant's ability to complete evaluations.
* History of seizures (excluding febrile seizures of childhood, or other isolated seizure episodes that were not due to epilepsy in the judgment of the Investigator, and required at most time-limited anticonvulsant treatment, and which occurred more than 7 years prior to the screening visit).
* Women who are pregnant or intend to become pregnant during the conduct of this study.
* Women who are nursing infants or intend to nurse infants during the conduct of this study.
* Known (or prior) hypersensitivity to donanemab, RG6289, or any excipients of RG6289.
* History of or active inflammatory bowel disease (e.g., Crohn disease or ulcerative colitis).
* Medical history of malignancy in the past 5 years, with the following exceptions:

  1. If considered to be cured or,
  2. If not being actively treated with anti-cancer therapy or radiotherapy and, in the opinion of the Investigator, is not likely to require treatment in the ensuing 5 years and,
  3. For prostate cancer or basal cell carcinoma, no significant progression over the previous 2 years.
  4. In-situ cervix carcinoma that has been successfully treated.
  5. Fully excised non-melanoma skin cancers or in-situ melanoma.
* Any surgery or hospitalization during the 4 weeks prior to screening or pre-planned/scheduled during the study period that, in the opinion of the Investigator, may compromise eligibility to the study. The Medical Monitor is available to the Investigator to advise and answer any questions.
* Inability to tolerate MRI procedures or contraindication to MRI, including, but not limited to, presence of pacemakers not compatible with MRI, aneurysm clips, artificial heart valves, ear implants, or foreign metal objects in the eyes, skin, or body that would contraindicate an MRI scan, or any other clinical history or examination finding that, in the judgment of the Investigator, would pose a potential hazard in combination with MRI
* Prior participation in an anti-amyloid therapy trial is allowed if it has been at least 1 year since the last study dose.
* Any other investigational treatment, including anti-amyloid small molecules (i.e., BACEi and GSIs, other GSMs) within five half-lives or 16 weeks prior to screening (calculated from the last safety follow-up visit of the previous study), whichever is longer. Note: The participant may be eligible for this study if it can be documented that he/she was randomized to placebo

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2030-06-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
Part 1: Change in amyloid load as measured by centiloid (CL) [F18]Florbetapir-PET as biomarker endpoint | Part 1: Screening, Month 9, and Month 18
  Evaluate the efficacy and safety of donanemab on change in amyloid load as measured by centiloid (CL) [F18] Florbetapir-PET in presenilin 1 (PSEN1) E280A mutation carriers (Part 1). CL calculated using [f18] Florbetapir PET non-partial volume corrected (regional spread function) standardized uptake value ratio cortical composite (F18 Florbetapir PET SUVR).
Part 2: Maintenance of Low Levels of Brain Amyloid as Measured by centiloid (Cl) [F18]Florbetapir-PET Following Combined Intervention of Donanemab and RG6289 | Duration of Part 2 Participation (up to 18 months)
  Evaluate the individual and relative efficacy and safety, as well as potential synergy, of donanemab, RG6289, and the combination of RG6289 with donanemab, to achieve and/or maintain low levels of brain amyloid as measured by centiloid (CL) [F18] Florbetapir-PET in asymptomatic and symptomatic PSEN1 E280A mutation carriers. CL calculated using [F18] Florbetapir-PET non-partial volume corrected (regional spread function) standardized uptake value ratio cortical composite (F18 Florbetapir-PET SUVR)

OTHER OUTCOMES:
Cerebrospinal Fluid Amyloid, TAU, and Other Biomarker Endpoints | Total duration of study participation (Up to 27 months)
  Change from baseline in cerebrospinal fluid (CSF) biomarkers including Aβ1-42, Aβ1-40, Aβ1-37, Aβ1-38, alpha-synuclein, GFAP, neurogranin, neurofilament light (NfL), pTau217, sTREM2, total tau, and YKL-40. Each resulting value will allow for the determination of Amyloid, TAU, and other protein trajectories related to Alzheimer's Disease Dementia. While each assay will have their own unit of measurement, each test will allow for comparison and confirmation of the presence and amount of targeted markers.
Plasma Amyloid, TAU, and Other Biomarker Endpoints | Total duration of study participation (Up to 27 months)
  Change from baseline in plasma biomarkers, including Aβ1-42, Aβ1-40, Aβ1-37, Aβ1-38, GFAP, NfL, pTau217, sTREM2, and YKL-4. Each resulting value will allow for the determination of Amyloid, TAU, and other protein trajectories related to Alzheimer's Disease Dementia within blood plasma. Each assay will have their own unit of measurement, and will allow for comparison and confirmation of the presence and amount of targeted markers.
Magnetic Resonance Imaging - Volumetric Measurements | Total duration of study participation (Up to 27 months)
  Change from baseline in volumetric magnetic resonance imaging (MRI) measures including whole brain volume, ventricular volume, entorhinal cortex volume, hippocampal volume, and temporal lobe volume.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Alexander, M.D., Principal Investigator — Banner Alzheimer's Institute; Jessica Langbaum, Ph.D., Principal Investigator — Banner Alzheimer's Institute; Eric Reiman, M.D., Principal Investigator — Banner Alzheimer's Institute; Yakeel T. Quiroz-Gaviria, Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Neurosciences Group of Antioquia, University of Antioquia, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: Yes